CLINICAL TRIAL: NCT06343259
Title: Comparison of The Effects of General Anesthesia and Spinal Anesthesia on The Development of Postoperative Myocardial Injury in Elderly Patients Undergoing Hip Surgery
Brief Title: The Effects of General Versus Spinal Anesthesia on Postoperative Myocardial Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Bilgehan Ayik, principal investigator, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2534
Record Dates: First submitted 2024-03-12; First posted 2024-04-02 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Myocardial Injury After Non-cardiac Surgery; Hypotension During Surgery; Anesthesia, General; Anesthesia, Spinal
Keywords: MINS; Anesthesia, General; Anesthesia, Spinal; Hip Fractures; Myocardial Infarction; Troponin T
MeSH Terms: conditions — Hip Fractures; Myocardial Infarction | interventions — Anesthesia, General; Propofol; Fentanyl; Rocuronium; Respiration, Artificial; Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (Active Comparator): After preoxygenation, intravenous fentanyl (1 μg/kg), propofol (2 mg/kg), and rocuronium (0.6 mg/kg) will be used for anesthesia induction. Intubation will be performed with a 7.0-8.0 sized tube, followed by the initiation of mechanical ventilation (tidal volume: 6-8 ml/kg, respiratory rate: 12 breaths/min). Sevoflurane will be used to maintain anesthesia (0.7-1 MAC), and remifentanil infusion will be administered for analgesia. Postoperatively, tramadol (1 mg/kg) and paracetamol (10 mg/kg) will be administered intravenously. Neuromuscular blockade will be reversed using sugammadex. Patients with an Aldrete Recovery Score ≥9 will be transferred to the post-anesthesia care unit after extubation.
  Interventions: Procedure: General Anesthesia
- Spinal Anesthesia (Active Comparator): Patients will be positioned laterally with the hip to be operated on the lower side, and skin asepsis will be ensured, followed by sterile draping. A dural puncture will be performed at the L3-4 spinal level using a 22-25 gauge Quincke-tip spinal needle. After the detection of cerebrospinal fluid, 7.5 mg of 0.5% hyperbaric bupivacaine will be slowly injected. Following a 10-minute interval, the sensory block level will be assessed using the pinprick test and modified Bromage scale, aiming for a T10 sensory block. Surgery will commence upon achieving adequate sensory block. Postoperatively, patients will be transferred to the recovery room. Patients failing to attain sufficient sensory block and experiencing pain will undergo transition to general anesthesia, terminating their cases.
  Interventions: Procedure: Spinal Anesthesia

INTERVENTIONS:
Procedure: General Anesthesia — After preoxygenation, intravenous fentanyl (1 μg/kg), propofol (2 mg/kg), and rocuronium (0.6 mg/kg) will be used for anesthesia induction. Intubation will be performed with a 7.0-8.0 sized tube, followed by the initiation of mechanical ventilation (tidal volume: 6-8 ml/kg, respiratory rate: 12 breaths/min). Sevoflurane will be used to maintain anesthesia (0.7-1 MAC), and remifentanil infusion will be administered for analgesia. Postoperatively, tramadol (1 mg/kg) and paracetamol (10 mg/kg) will be administered intravenously. Neuromuscular blockade will be reversed using sugammadex. Patients with an Aldrete Recovery Score ≥9 will be transferred to the post-anesthesia care unit after extubation.
  Other Names: propofol; fentanyl; rocuronium; sevoflorane; mechanical ventilation
  Arms: General Anesthesia
Procedure: Spinal Anesthesia — Patients will be positioned laterally with the hip to be operated on the lower side, and skin asepsis will be ensured, followed by sterile draping. A dural puncture will be performed at the L3-4 spinal level using a 22-25 gauge Quincke-tip spinal needle. After the detection of cerebrospinal fluid, 7.5 mg of 0.5% hyperbaric bupivacaine will be slowly injected. Following a 10-minute interval, the sensory block level will be assessed using the pinprick test and modified Bromage scale, aiming for a T10 sensory block. Surgery will commence upon achieving adequate sensory block. Postoperatively, patients will be transferred to the recovery room. Patients failing to attain sufficient sensory block and experiencing pain will undergo transition to general anesthesia, terminating their cases.
  Other Names: bupivacain
  Arms: Spinal Anesthesia

SUMMARY:
In this prospective, randomized, single-blind study, we aim to compare the effects of general anesthesia and spinal anesthesia on postoperative myocardial injury in elderly patients undergoing hip surgery. Cardiovascular events are a leading cause of mortality and morbidity following non-cardiac surgery, with myocardial injury after non-cardiac surgery (MINS) being a significant concern. MINS, characterized by asymptomatic elevation of troponin levels without accompanying ECG findings, is closely associated with postoperative mortality. With the increasing prevalence of comorbidities in the elderly population and the rising frequency of non-cardiac surgeries in this demographic, understanding the effects of different anesthesia types on postoperative myocardial injury is crucial.

DETAILED DESCRIPTION:
Cardiovascular events constitute the leading cause of mortality and morbidity following non-cardiac surgery. Myocardial Injury after Non-cardiac Surgery (MINS) is a condition diagnosed postoperatively characterized by asymptomatic troponin elevation alone. Distinguishing it from myocardial infarction, it lacks symptoms and concurrent Electrocardiography (ECG) findings, yet it correlates closely with postoperative mortality. Detection can be facilitated through troponin monitoring from preoperative period to up to 72 hours postoperatively.

The Vascular Events in Noncardiac Surgery Patient Cohort Assessment (VISION) study, designed to evaluate major vascular events in patients undergoing non-cardiac surgery, reported a global prevalence of MINS at 8% with over a threefold increase in 30-day mortality. The diagnostic threshold for MINS as determined by the VISION study is a non-Hs troponin T level of ≥0.03 ng/mL.

With the increasing elderly population burdened with comorbidities globally, the frequency of non-cardiac surgeries in elderly patients has risen. Despite advancements in surgical and anesthetic fields, the incidence of MINS and associated mortality continue to escalate. Risk factors associated with MINS highlight age over 75 and the presence of comorbidities. Orthopedic surgeries are most commonly performed in elderly patients, with perioperative acute myocardial infarction (MI) incidence shown to increase by 31-fold in knee surgeries and 25-fold in hip surgeries. Postoperative pain and opioid use in this patient group significantly contribute to overlooked myocardial ischemia.

In a sub-study of the VISION trial examining cardiovascular outcomes of orthopedic surgery, the incidence of MINS was reported at 11.9%, with 30-day mortality rates of 1% in MINS-absent patients and 9.8% in MINS-present patients, markedly higher than non-orthopedic surgeries.

Several studies have identified perioperative and postoperative hypotension as the primary risk factor for MINS, emphasizing the importance of anesthesia management in preventing perioperative hypotension. However, no study has specifically focused on the relationship between chosen anesthesia technique and the development of hypotension and MINS. George R. and colleagues conducted a prospective observational cohort study in India analyzing the incidence and risk factors of MINS, finding a higher incidence in patients receiving peripheral nerve blocks compared to general anesthesia and spinal anesthesia, particularly in patients with high cardiac comorbidities. Nonetheless, no significant relationship was observed between the chosen anesthesia technique and the development of MINS in the orthopedic surgery subgroup of the VISION study.

In this prospective, randomized, single-blind study, we aim to compare the effects of general anesthesia and spinal anesthesia on postoperative myocardial injury in elderly patients undergoing hip surgery.

ELIGIBILITY:
Inclusion Criteria:

* who will undergo hip surgery
* ASAII-III
* Over the age of 65

Exclusion Criteria:

* Patients diagnosed with sepsis, pulmonary embolism, decompensated heart failure, chronic kidney failure.
* Patients who underwent cardioversion in the last 6 months or experienced myocardial infarction.
* Patients with a surgical history in the last month.
* Patients who required intubation in the intensive care unit.
* Patients with a baseline Hs-Troponin T value exceeding 20 ng/L.
* Patients with a postoperative peak Hs-Troponin T value higher than baseline.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2024-08-05 (Estimated); Study Completion 2024-08-18 (Estimated)

PRIMARY OUTCOMES:
Myocardial Injury After Non-Cardiac Surgery (MINS) | up to 72 hour
  Blood samples for hs-Troponin T values were obtained at 0 hours in the recovery room, followed by assessments at 6, 12, 24, 48, and 72 hours either in the ward or in the intensive care unit.The baseline values were within the normal range, with postoperative hsTnT measurements ranging between 20 and 65 ng/L, and those with at least a 5 ng/L absolute change or hsTnT levels of 65 ng/L and above were considered as MINS.

SECONDARY OUTCOMES:
The duration of intensive care unit (ICU) stay | up to 90 days
  The intensive care unit (ICU) stay durations of patients who develop MINS and those who do not develop MINS will be recorded and compared.
The duration of hospital stay | up to 90 days
  The hospital stay durations of patients who develop MINS and those who do not develop MINS will be recorded and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No